CLINICAL TRIAL: NCT05975593
Title: MicroEnvironment Tumor Effects of Radiotherapy - Comprehensive Radiobiology Assessment TRial (METEOR-CRATR)
Brief Title: MicroEnvironment Tumor Effects of Radiotherapy - Comprehensive Radiobiology Assessment TRial
Acronym: METEOR-CRATR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202307103; U54CA274318 (NIH)
Record Dates: First submitted 2023-07-24; First posted 2023-08-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Cervical Carcinoma; Locally Advanced Cervical Cancer; Locally Advanced Pancreas Cancer; Locally Advanced Pancreatic Carcinoma; Locally Advanced Pancreatic Cancer; Cervical Cancer; Pancreas Cancer; Pancreatic Cancer; Cancer of the Cervix; Cancer of the Pancreas
Keywords: Radiotherapy; Chemotherapy; Cervical cancer; Pancreatic cancer; Biospecimen
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pancreatic Neoplasms | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: 30 cervical cancer patients and 30 pancreatic cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cervical Cancer (Other): * Patients will have blood and tumor collected at various time points throughout participation in the study.
  * Patients will have standard of care imaging obtained at various time points and a diffusion basis spectrum imaging (DBSI) MRI will be obtained at the end of standard of care MRI.
  Interventions: Other: Tumor collection via biopsy; Other: Blood collection; Device: Diffusion basis spectrum imaging (DBSI) magnetic resonance imaging (MRI)
- Pancreatic Cancer (Other): * Patients will have blood and tumor collected at various time points throughout participation in the study.
  * Patients will have standard of care imaging obtained at various time points and a diffusion basis spectrum imaging (DBSI) MRI will be obtained at the end of standard of care MRI.
  Interventions: Other: Tumor collection via biopsy; Other: Blood collection; Device: Diffusion basis spectrum imaging (DBSI) magnetic resonance imaging (MRI)

INTERVENTIONS:
Other: Tumor collection via biopsy — Cervical cancer: Pre-radiation therapy, 1 week after beginning radiation therapy, 3 weeks after beginning radiation therapy, and recurrence.
  Pancreatic cancer: pre-stereotactic body radiotherapy, 12 weeks after completion of radiotherapy, and recurrence.
Other: Blood collection — Cervical cancer: pre-radiation therapy, 1 week after beginning radiation therapy, 3 weeks after beginning radiation therapy, 6 weeks after completing radiation therapy, 12 weeks after completing radiation therapy, and recurrence.
  Pancreatic cancer: pre-stereotactic body radiotherapy, 6 weeks after completion of radiotherapy, 12 weeks after completion of radiotherapy, surgery (if applicable), and recurrence
Device: Diffusion basis spectrum imaging (DBSI) magnetic resonance imaging (MRI) — Cervical cancer: initial staging, 12 weeks after completing radiation therapy, and recurrence.
  Pancreatic cancer: initial staging, stereotactic body radiotherapy (SBRT) simulation, 12 weeks after completing radiation therapy, and recurrence.
  The imaging will be performed when possible.
  Other Names: DBSI MRI

SUMMARY:
This study is a dynamically adjustable prospective longitudinal study designed to capture biospecimen (biopsy, blood, surgical) and multimodal treatment-related data (imaging, dosimetry, clinical) before, during, and after treatment with definitive-intent chemoradiotherapy for patients with locally advanced cervical and pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of intent to receive radiotherapy for one of the following diagnoses:

  * Cervical cancer
  * Pancreatic cancer
* ECOG performance status ≤ 2
* At least 18 years old
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Any issue (medical, anatomic, other) that might preclude safe acquisition of biospecimens at the discretion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in tumor microenvironment | From start of follow-up through completion of follow-up (estimated to be 5 years)
  Generalized linear mixed effects models will be first used to capture the changes in the longitudinal values of a single assay output over time for a given biospecimen. Random effects will be used to describe the correlation of repeated measures on the same subject over time.

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be presented at scientific meetings & published in journals. Individual-level & aggregate genomic data will be deposited/made available through GEO & SRA. Includes sequence, transcriptomic, epigenomic, & gene expression data. Raw mass spectra & unprocessed proteomic data will be shared through publisher mechanisms. Will use PRIDE & ProteomeEXchange to share protein identifications & spectral evidence. METEOR-BLST will collaborate with ROBIN centers to share expertise, data reporting and discovering of radiation biology. Data generated in this proposal will be shared with the scientific community subject to NIH & institutional regulations. BLST will manage & assist in dissemination of omics data generated. NIMS data will be deposited at MetaboLights. CODEX-based imaging data will be as supplemental files within manuscripts. Processed data will be available through CIELO. Model organisms generated will be distributed freely, or deposited into a repository/stock center.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting with the acceptance date of initial publication.
Access Criteria: Scientific progress and publications will be posted on the METEOR website. The respective departments of the PIs and co-Is also maintain web sites where information and links on the investigators' work are posted. The PIs and co-Is additionally have lab web sites where summaries of the scientific progress on projects and research interests are posted.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu